CLINICAL TRIAL: NCT01630057
Title: An Open-label, Randomized, Multi-centre, Superiority Study to Compare, in Patients With Partial Onset Seizures, the Efficacy and Safety of Adjunctive Zonisamide vs Replacement With Zonisamide of the Last Added Antiepileptic Drug
Brief Title: Evaluation of the Efficacy and Safety of Adjunctive Zonisamide vs Replacement With Zonisamide of the Last Added Antiepileptic Drug
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E2090-E039-401
Record Dates: First submitted 2010-11-16; First posted 2012-06-28 (Estimated); Last update posted 2014-07-14 (Estimated); Status verified 2014-07

CONDITIONS: Partial Seizures
MeSH Terms: conditions — Seizures | interventions — Replantation; Zonisamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Adjunctive Zonisamide (Experimental): Patients will be gradually down-titrated from the first add-on following a drug-specific scheme decided by the investigator. Discontinued from the first add-on, patients will remain on duotherapy until the end of the study, or until the clinical situation mandates withdrawal from the study, e.g. in case of seizure worsening or adverse events.
  Interventions: Drug: Adjunctive Zonisamide
- Replacement with Zonisamide (Active Comparator): Patients will continue to receive zonisamide as third drug
  Interventions: Drug: Replacement with Zonisamide

INTERVENTIONS:
Drug: Adjunctive Zonisamide — Patients will be gradually down-titrated from the first add-on following a drug-specific scheme decided by the investigator. Discontinued from the first add-on, patients will remain on duotherapy until the end of the study, or until the clinical situation mandates withdrawal from the study, e.g. in case of seizure worsening or adverse events.
  Arms: Adjunctive Zonisamide
Drug: Replacement with Zonisamide — Patients will continue to receive zonisamide as third drug
  Arms: Replacement with Zonisamide

SUMMARY:
An open-label, randomized, multi-centre, superiority study to assess that, in patients who respond to zonisamide added as third drug after failure of a two-drug combination therapy, the triple therapy is superior to the conversion to a double therapy including zonisamide.

ELIGIBILITY:
Patients with localization-related epilepsy, who have added a second drug to the monotherapy, haven't obtained an adequate reduction of seizure frequency with this combination and have responded to zonisamide added as third drug for at least three months.

Inclusion criteria:

* Age ≥ 18 years;
* Patients with non progressive localization-related epilepsy;
* Patients who are able and willing to give written Informed Consent;
* Current treatment with three antiepileptic drugs. The last antiepileptic drug introduced must be zonisamide;
* 50% or greater seizure reduction* as assessed after an at least three-month maintenance period with zonisamide.

  * = seizure frequency before starting zonisamide must be documented checking case histories.

Exclusion criteria:

* Patients contraindicated for zonisamide use (see SmPC);
* Patients with renal or hepatic impairment;
* Pregnant or lactating women;
* Women of childbearing age who are not willing to use any contraceptive method with established efficacy.
* Patients suffering from clinically significant psychiatric illness, psychological or behavioral problems which could interfere with study participation;
* Patients with a history (within the last 12 months) of alcohol or drug abuse or dependency;
* Patients who have been on an investigational drug or device within 30 days prior to the initiation of the present study;
* Patients with a documented computed axial tomography (CAT) scan or magnetic resonance imaging (MRI) scan confirming the presence of a progressive neurological lesion within 12 months of the screening visit.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2009-09; Primary Completion 2011-06 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability in patients who respond to zonisamide added as third drug after failure of a two-drug combination therapy | 13 months

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Striano, Principal Investigator — Federico II University
Locations (19):
- Italy (19):
  - UOC Neurofisiopatologia PO S. Salvatore, L’Aquila, Italy
  - AOU Ospedali riuniti Umberto I -G.M Lancisi-G.Salesi, Ancona
  - AO Universitaria Consorziale Policlinico di Bari, Bari
  - Irccs "E. Medea", Bosisio Parini
  - Struttura di Neurofisiopatologia, Universit? degli studi di Cagliari, Cagliari
  - IRCCS "Eugenio Medea" Polo Scientifico di Conegliano, Conegliano
  - AOU di Ferrara Arcispedale S. Anna, Ferrara
  - Presidio Ospedale "S.Antonio Abate di Gallarate", Gallarate
  - AO della Provincia di Lodi, Lodi
  - IRCCS Centro neurolesi "Bonino Pulejo" di Messina, Messina
  - AO di Rilievo Nazionale Antonio Cardarelli, Napoli
  - AO Universitaria Federico II, Napoli
  - AO Universitaria Policlinico Paolo Giaccone dell'Universit? degli Studi di Palermo, Palermo
  - AO Universitaria -Pisana, Pisa
  - AO Regionale "San Carlo" di Potenza, Potenza
  - PO "Misericordia e dolce"-USL 4 di Prato, Prato
  - Azienda Complesso Ospedaliero San Filippo Neri, Roma
  - Umberto I Policlinico di Roma, Roma
  - Ospedale SS Giovanni e Paolo Azienda ULSS 12 Veneziana, Venezia